CLINICAL TRIAL: NCT04030910
Title: 'LIFEView' Audiovisual Technology: Virtual Travel to Support Wellbeing and Quality of Life at the End of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Bruyere Continuing Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LIFEView 2
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Palliative Care; Terminal Illness; Quality of Life; Psychological Distress
Keywords: Life review; Reminiscence; Technology; Existential distress; Virtual travel; Well-being

STUDY DESIGN:
Intervention Model Description: All eligible patients will be recruited to receive the intervention ("LIFEView").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 'LIFEView' intervention (Experimental): The 'LIFEView' session(s) involves the use of audiovisual software by Motitech AS (technology provided by and used with permission from Motitech AS). For its primary uses as Motiview, the audiovisual software was coupled to a mobile user-adapted cycle-trainer. Since a secondary benefit of the virtual cycle trip may include reminiscence which may in-turn facilitate conversation of past experiences, the audiovisual software is being adapted for use in reminiscence therapy for a palliative care population.
  As there is an extensive library available to participants and 'LIFEView' sessions could potentially be longer than feasible for research personnel to conduct, each 'LIFEView' session will be limited to up to 3 videos per session or up to 1 hour of videos per session, whichever is a shorter duration. Additional post-study 'LIFEView' sessions can be provided upon request from participants.
  Interventions: Other: 'LIFEView'

INTERVENTIONS:
Other: 'LIFEView' — A prototype audiovisual technology in development by Motitech AS.

SUMMARY:
This study is looking to assess the use of an audio-video technology called 'LIFEView' using a laptop and large-screen TV. This tool intends to support life review or reminiscence of past experiences, escape from current surroundings using virtual travel, or virtual visits to a location that one might have liked to visit in their lifetime but could not. We hope that by using this technology, we can support better wellbeing and quality of life for patients receiving palliative care services within the community and on an inpatient palliative care unit, or for patients at the end-of-life within Bruyère long-term care homes.

Due to the potential for disorientation and reduced physical mobility, patients receiving palliative and end-of-life care may be unable to fully enjoy an immersive experience using a virtual reality (VR) headset. To reduce the possibility of disorientation that may arise from using a VR headset with 'LIFEView', our research team will use the 'LIFEView' prototype software loaded on a laptop and connected to a mobile high-definition 50" TV for inpatient PCU and LTC facility use, or to a patient's personal TV within their residence in the community. This setup will also improve accessibility to 'LIFEView' as a result of its relatively low-tech requirements (i.e. TV + laptop), and allows for an opportunity for patients and their loved ones to share cherished memories and stories.

DETAILED DESCRIPTION:
This project is designed to address the psychosocial and existential suffering commonly experienced by palliative care patients. Technology-based reminiscence and dignity therapy interventions have been demonstrated to improve well-being and quality of life in older adults (Lazar et al, 2014), although little evidence exists to support the use of these technology-based interventions in a palliative care context.

These technologies may require modification to meet the needs of PEOLC patients that are at risk for delirium, a neuropsychiatric condition characterized by fluctuating disruptions in awareness, focus and cognition (American Psychiatric Association, 2013). Delirium can be experienced by up to 88% of patients at the end of life (Hosie et al., 2013). Moreover, patients in PEOLC settings may also have limited mobility or may be bedbound. Due to the potential for disorientation and reduced physical mobility, patients receiving PEOLC may be unable to fully enjoy an immersive experience using a virtual reality (VR) headset. To reduce the possibility of disorientation that may arise from using a VR headset with 'LIFEView', our research team plans to use the 'LIFEView' prototype software loaded on a laptop and connected to a mobile high-definition 40-42" TV for inpatient PCU and LTC facility use, or to a patient's personal TV within their residence in the community.

ELIGIBILITY:
Inclusion Criteria:

• Any patients who are able to complete the outcome measures (Section 5.0 Outcomes) and capable of consenting to participating in the research study will be included.

Exclusion Criteria:

Patients experiencing the following, as determined by the clinical care team:

* Delirium
* Severe cognitive impairment (as determined by the clinical care team)
* Known behavioural abnormalities (e.g. overtly aggressive behavior) that in the opinion of the clinical care team might impede any meaningful participation in the project
* A score of <30% on the Palliative Performance Scale (PPS) (Anderson et al., 1996) at the time of consent
* Individuals who are already currently using Motiview paired with a exercise bicycle in the LTC setting
* Those who are in the opinion of attending physician or clinical team too unwell to participate in the project
* Unable to complete outcome measures indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in psychological and physical symptoms measured by the Edmonton Symptom Assessment System-revised (ESAS-r) (Bruera et al., 1991; Watanabe et al., 2011) | At least 24 hours before using 'LIFEView', and directly after and 48 hours after using 'LIFEView' (pre- and post-'LIFEView')
  The ESAS-r is a 9-item symptom assessment tool that assesses pain, tiredness, drowsiness, nausea, lack of appetite, shortness of breath, depression, anxiety, and feeling of wellbeing. Each item is rated by patients on a 0-10 scale (0= best possible, 10= worst possible).

SECONDARY OUTCOMES:
Change in quality of life measured by the McGill Quality of Life-Revised questionnaire (Cohen et al., 2017) | At least 24 hours before using 'LIFEView', and 48 hours after using 'LIFEView' (pre- and post-'LIFEView')
  The MQOL-R will be used to assess patient quality of life. There are 4 parts to the questionnaire on overall quality of life, physical symptoms, feelings and thoughts, and social aspects of the participant's life. Each statement is rated on a 0-10 scale (0= worst possible,10= best possible).
Psychosocial effects and aspects of quality of life as determined by semi-structured interviews for consenting participants and their consenting family member(s) or caregiver(s). | Within 24 hours of using 'LIFEView' (post-'LIFEView')
  These interviews will explore the impact of the 'LIFEView' intervention on patient quality of life, patient-family and patient-caregiver interactions, perceptions of the 'LIFEView' intervention as a tool to improve well-being and quality of life in palliative care settings, and feasibility of using volunteer services to support the long-term sustainability of this intervention across care settings.
Change in heart rate | At least 24 hours before using 'LIFEView', and directly after using 'LIFEView' (pre- and post-'LIFEView')
  Heart rate (beats per minute; bpm) will be measured using a wireless cuff.
Change in blood pressure | At least 24 hours before using 'LIFEView', and directly after using 'LIFEView' (pre- and post-'LIFEView')
  Blood pressure (mm Hg) will be measured using a wireless cuff.

OTHER OUTCOMES:
Aspects of participant's level of general well-being as per the Greater Cincinnati Chapter Well-Being Observation tool (Rentz, 2002; Kinney & Rentz, 2005) during the 'LIFEView' session, and other observable phenomena | From initiation of the 'LIFEView' session and directly after using 'LIFEView' (during and post-'LIFEView')
  The Greater Cincinnati Chapter Well-Being Observation tool will be used by the research team members to assess each patient's state of general well-being. There are 6 domains, for which each statement is rated on a 0-4 scale (0= never, 1= rarely, 2= some of the time, 3= most of the time, 4= always).
  Observational field notes will be taken by the Research Coordinator during the course of study participation on observable phenomena before, during, and after the 'LIFEView' session (e.g. verbalized reminiscence, feelings… etc.). Patients and their family members will only be identified by their participant study ID in field notes.

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Hackbusch, Principal Investigator — Bruyère Continuing Care; Jill Rice, MD, CCFP(PC), Principal Investigator — Bruyère Continuing Care
Locations (1):
- Bruyere Continuing Care, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CW, Chow AY, Chan CL. The effects of life review interventions on spiritual well-being, psychological distress, and quality of life in patients with terminal or advanced cancer: A systematic review and meta-analysis of randomized controlled trials. Palliat Med. 2017 Dec;31(10):883-894. doi: 10.1177/0269216317705101. Epub 2017 May 10. PMID 28488923
- [Background] Ando M, Tsuda A, Morita T. Life review interviews on the spiritual well-being of terminally ill cancer patients. Support Care Cancer. 2007 Feb;15(2):225-31. doi: 10.1007/s00520-006-0121-y. Epub 2006 Sep 12. PMID 16967303
- [Background] Warth M, Kessler J, Koehler F, Aguilar-Raab C, Bardenheuer HJ, Ditzen B. Brief psychosocial interventions improve quality of life of patients receiving palliative care: A systematic review and meta-analysis. Palliat Med. 2019 Mar;33(3):332-345. doi: 10.1177/0269216318818011. Epub 2019 Jan 16. No abstract available. PMID 30648926
- [Background] Lazar A, Thompson H, Demiris G. A systematic review of the use of technology for reminiscence therapy. Health Educ Behav. 2014 Oct;41(1 Suppl):51S-61S. doi: 10.1177/1090198114537067. PMID 25274711
- [Background] Hosie A, Davidson PM, Agar M, Sanderson CR, Phillips J. Delirium prevalence, incidence, and implications for screening in specialist palliative care inpatient settings: a systematic review. Palliat Med. 2013 Jun;27(6):486-98. doi: 10.1177/0269216312457214. Epub 2012 Sep 17. PMID 22988044
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Watanabe SM, Nekolaichuk C, Beaumont C, Johnson L, Myers J, Strasser F. A multicenter study comparing two numerical versions of the Edmonton Symptom Assessment System in palliative care patients. J Pain Symptom Manage. 2011 Feb;41(2):456-68. doi: 10.1016/j.jpainsymman.2010.04.020. Epub 2010 Sep 15. PMID 20832987
- [Background] Kinney JM, Rentz CA. Observed well-being among individuals with dementia: Memories in the Making, an art program, versus other structured activity. Am J Alzheimers Dis Other Demen. 2005 Jul-Aug;20(4):220-7. doi: 10.1177/153331750502000406. PMID 16136845
- [Background] Anderson F, Downing GM, Hill J, Casorso L, Lerch N. Palliative performance scale (PPS): a new tool. J Palliat Care. 1996 Spring;12(1):5-11. PMID 8857241
- [Background] Lee JS, Hurley MJ, Carew D, Fisher R, Kiss A, Drummond N. A randomized clinical trial to assess the impact on an emergency response system on anxiety and health care use among older emergency patients after a fall. Acad Emerg Med. 2007 Apr;14(4):301-8. doi: 10.1197/j.aem.2006.11.017. Epub 2007 Mar 1. PMID 17331915
- [Background] Stromgren AS, Goldschmidt D, Groenvold M, Petersen MA, Jensen PT, Pedersen L, Hoermann L, Helleberg C, Sjogren P. Self-assessment in cancer patients referred to palliative care: a study of feasibility and symptom epidemiology. Cancer. 2002 Jan 15;94(2):512-20. doi: 10.1002/cncr.10222. PMID 11900236
- [Background] Bernard H. Research Methods in Anthropology: Qualitative and Quantitative Approaches. 2nd ed. Thousand Oaks, CA: Sage Publications; 1995 1995.
- [Background] Patton M. Qualitative Research and Evaluation Methods. 4th ed. Thousand Oaks, CA: Sage Publications, Inc; 2015.
- [Background] Guest G, Bunce A, Johnson L. How Many Interviews Are Enough ? An Experiment with Data Saturation and Variability. Fam Heal Int 2006;18(1):59-82 doi:10.1177/1525822X05279903.
- [Background] Mitchell AJ, Meader N, Symonds P. Diagnostic validity of the Hospital Anxiety and Depression Scale (HADS) in cancer and palliative settings: a meta-analysis. J Affect Disord. 2010 Nov;126(3):335-48. doi: 10.1016/j.jad.2010.01.067. Epub 2010 Mar 5. PMID 20207007
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Hickey G, Kipping C. A multi-stage approach to the coding of data from open-ended questions. Nurse Res. 1996 Oct 1;4(1):81-91. doi: 10.7748/nr.4.1.81.s9. PMID 27707369
- [Background] Rentz CA. Memories in the making: outcome-based evaluation of an art program for individuals with dementing illnesses. Am J Alzheimers Dis Other Demen. 2002 May-Jun;17(3):175-81. doi: 10.1177/153331750201700310. PMID 12083348
- [Background] American Psychiatric Association. Delirium due to a general medical condition. Diagnostic and Statistical Manual of Mental Disorders, Fifth edition (DSM-5). Arlington, VA: American Psychiatric Association; 2013. p. 596-602.
- [Background] Bedard G, Zeng L, Zhang L, Lauzon N, Holden L, Tsao M, Danjoux C, Barnes E, Sahgal A, Poon M, Chow E. Minimal clinically important differences in the Edmonton symptom assessment system in patients with advanced cancer. J Pain Symptom Manage. 2013 Aug;46(2):192-200. doi: 10.1016/j.jpainsymman.2012.07.022. Epub 2012 Nov 22. PMID 23177724
- [Background] Mercadante S, Adile C, Lanzetta G, Mystakidou K, Maltoni M, Guilherme Soares L, De Santis S, Ferrera P, Valenti M, Rosati M, Rossi R, Cortegiani A, Masedu F, Marinangeli F, Aielli F. Personalized Symptom Goals and Patient Global Impression on Clinical Changes in Advanced Cancer Patients. Oncologist. 2019 Feb;24(2):239-246. doi: 10.1634/theoncologist.2017-0668. Epub 2018 May 16. PMID 29769382
- [Background] Hui D, Bruera E. Minimal clinically important differences in the edmonton symptom assessment system: the anchor is key. J Pain Symptom Manage. 2013 Mar;45(3):e4-5. doi: 10.1016/j.jpainsymman.2012.12.003. No abstract available. PMID 23465763
- [Background] Hui D, Shamieh O, Paiva CE, Khamash O, Perez-Cruz PE, Kwon JH, Muckaden MA, Park M, Arthur J, Bruera E. Minimal Clinically Important Difference in the Physical, Emotional, and Total Symptom Distress Scores of the Edmonton Symptom Assessment System. J Pain Symptom Manage. 2016 Feb;51(2):262-9. doi: 10.1016/j.jpainsymman.2015.10.004. Epub 2015 Oct 19. PMID 26482223